CLINICAL TRIAL: NCT01059994
Title: Role of Skeletal Muscle Nitric Oxide Production in Age-related Fatigue and Fatigability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-213
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2018-11

CONDITIONS: Fatigue; Aging
Keywords: fatigue; aging
MeSH Terms: conditions — Fatigue | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo sildenafil young (Placebo Comparator): Younger subjects (ages 20-35) were administered placebo sildenafil orally daily for 1 week.
  Interventions: Drug: Placebo sildenafil
- sildenafil young (Experimental): Younger subjects (ages 20 -35) were administered sildenafil daily (25 mg/day) orally for 1 week.
  Interventions: Drug: Sildenafil
- placebo sildenafil older (Placebo Comparator): Older subjects (ages 60-80) were administered placebo sildenafil orally daily for 1 week.
  Interventions: Drug: Placebo sildenafil
- sildenafil older (Experimental): Older subjects (ages 60 - 80) were administered sildenafil daily (25 mg/day) orally for 1 week.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Placebo sildenafil — Oral, daily, 1 week.
  Other Names: Viagra
  Arms: placebo sildenafil older; placebo sildenafil young
Drug: Sildenafil — oral, 25mg, daily for 1 week
  Other Names: Viagra
  Arms: sildenafil older; sildenafil young

SUMMARY:
This is a pilot study funded by the National Institutes of Health. In this project, we will investigate the potential effect of skeletal muscle nitric oxide (NO) production on muscle strength and physical function in older individuals. We propose to test a new method that may enable simultaneous determination of both vascular and skeletal muscle NO production for the first time in humans. Further, we will determine whether augmentation of NO-mediated responses, by administration of sildenafil citrate (Viagra), reduces fatigue and fatigability in older individuals.

DETAILED DESCRIPTION:
Fatigue is highly prevalent and associated with future mortality in older individuals. Even in non-disabled older persons, fatigue may be the primary reason for activity limitation. However, understanding the etiology of fatigue in this population has been hampered by differing or imprecise definitions of fatigue. As a result, the term fatigue has been proposed to refer to the subjective experience of tiredness or lack of energy, whereas the term fatigability should refer to the susceptibility to fatigue induced by activity of any kind (mental, physical, etc). Skeletal muscle activity can contribute to the perception of overall fatigue as well as produce a type of localized fatigue within skeletal muscle. Skeletal muscle fatigue is defined as a decline in skeletal muscle performance resulting from muscle activity.

We hypothesize that skeletal muscle NO-mediated responses are reduced with aging due to decreased skeletal muscle NO production. NO is well-known to elicit vasodilation through stimulation of cGMP signaling, and NO-mediated changes in muscle perfusion may influence both skeletal muscle and overall fatigue. To measure skeletal muscle NO production, we will infuse a stable isotope tracer of arginine, the precursor of NO, and measure its conversion across the leg and in skeletal muscle to citrulline (which is another product of the reaction that produces NO). If successful, this method will allow the study of relative changes in vascular and muscle NO production that occur with aging and other conditions (e.g., hypertension, Duchenne muscular dystrophy). We will also determine whether age-related differences in muscle perfusion and NO-cGMP signaling exist between younger and older groups. As impaired redox homeostasis and ryanodine receptor S-nitrosylation and phosphorylation have been implicated in skeletal muscle fatigue, we will assess skeletal muscle redox homeostasis and ryanodine receptor S-nitrosylation in these experiments. We hypothesize that aging will shift muscle redox homeostasis to a more oxidized state.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20-35 yrs, and 60-80 yrs.
* 2. Ability to sign consent form (score >23 on the 30-item Mini Mental State Examination, MMSE)
* 3. Stable body weight for at least 3 months

Exclusion Criteria:

* 1. Physical dependence or frailty (impairment in any of the Activities of Daily Living (ADL), history of falls (>2/year) or significant weight loss in the past year)
* 2. Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
* 3. Pregnancy
* 4. Significant heart, liver, kidney, blood or respiratory disease
* 5. Peripheral vascular disease
* 6. Diabetes mellitus or other untreated endocrine disease
* 7. Active cancer
* 8. Use of nitrates
* 9. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
* 10. Alcohol or drug abuse
* 11. Severe depression (>5 on the 15-item Geriatric Depression Scale, GDS)
* 12. Cardiac abnormalities such as a cardiac shunt or previously diagnosed pulmonary hypertension.
* 13. Systolic blood pressure <100 or >150, diastolic blood pressure <60 or >90.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Durham, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males in the age groups of 20-35 and 60-80 were recruited. Subjects were screened and enrolled at the University of Texas Medical Branch in the Institute for Translational Sciences Clinical Research Center (ITS-CRC).
Pre-assignment Details: Participants who failed screening, did not otherwise meet inclusion criteria, or decided not to participate were excluded before being assigned to intervention groups.
Groups:
- Sildenafil Placebo Young; Sildenafil Placebo Older: Sildenafil placebo: Oral, daily, 1 week.
Period: Overall Study
Arm/Group | Sildenafil Placebo Young | Sildenafil Young | Sildenafil Placebo Older | Sildenafil Older
Started | 3 | 2 | 3 | 4
Completed | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Sildenafil Young; Placebo Sildenafil Older: Sildenafil placebo: Oral, daily, 1 week.
- Total: Total of all reporting groups
Arm/Group | Placebo Sildenafil Young | Sildenafil Young | Placebo Sildenafil Older | Sildenafil Older | Total
Number analyzed (Participants) | 3 | 2 | 3 | 4 | 12
Age, Customized [Mean (Standard Deviation); unit: years] | 25 (6) | 29 (4) | 63 (5) | 74 (4) | 51 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 2 | 3 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Fatigue After 1 Week of Placebo or Sildenafil
Description: Muscle fatigue was tested before and after 1 week of placebo/sildenafil (25mg/day) treatment.
  Subjects were asked to perform maximum effort isokinetic knee extensions until force production reached 50% of their MVC (maximum voluntary contraction). Data was collected as number of successful repetitions completed between start and 50% MVC.
  Data is presented as percent change in repetitions (1 week of treatment / baseline).
Time Frame: baseline to 1 week
Measure: Mean (Standard Deviation); unit: percent change of successful repetitions
Arm/Group | Placebo Sildenafil Young | Sildenafil Young | Placebo Sildenafil Older | Sildenafil Older
Number analyzed (Participants) | 3 | 2 | 3 | 3
percent change of successful repetitions | 107 (5) | 115 (10) | 54 (31) | 158 (27)
Statistical Analysis 1: Comparison: Placebo Sildenafil Young vs Sildenafil Young; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Protein Synthesis Rate After 1 Week of Sildenafil or Placebo
Description: Skeletal muscle protein synthesis, measured as the fractional synthesis rate (the percent of the total synthesized per unit time) after 1 week of either Placebo or Sildenafil (25 mg/day). Example: if FSR = 0.06 hr-1 it means that 6% of proteins in a given sample were synthesized in the last hour or proteins is synthesized at 6% per hour. A higher rate means that more synthesis is occurring.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: fraction of proteins synthesized/hr
Arm/Group | Placebo Sildenafil Young | Sildenafil Young | Placebo Sildenafil Older | Sildenafil Older
Number analyzed (Participants) | 3 | 2 | 3 | 3
fraction of proteins synthesized/hr | 0.06 (0.03) | 0.11 (0.04) | 0.04 (0.01) | 0.10 (0.03)
Statistical Analysis 1: Comparison: Placebo Sildenafil Young vs Sildenafil Young; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo Sildenafil Young | Sildenafil Young | Placebo Sildenafil Older | Sildenafil Older
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes